CLINICAL TRIAL: NCT05735067
Title: The Impact of Body Weight on Clinical and Immunological Outcomes in Relapse-Remitting Multiple Sclerosis Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: German University in Cairo (Other)
Responsible Party: Principal Investigator, Mohamed Youssef Elsayed, Research assistant in Clinical Pharmacology and Pharmacogenomics Research Gruop, German University in Cairo
Other Study IDs: MSINF
Record Dates: First submitted 2023-02-09; First posted 2023-02-21 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis, IFB 1a
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: RRMS patients who received Interferon beta 1a and have normal weight
  Interventions: Other: Blood sample collection
- Group 2: RRMS patients who received Interferon beta 1a and have are obese
  Interventions: Other: Blood sample collection

INTERVENTIONS:
Other: Blood sample collection — 5 ml of blood samples were withdrawn from RRMS patients

SUMMARY:
Our study aimed to investigate the effect of interferon beta 1a on the clinical and immunological parameters in Egyptian relapse-remitting multiple sclerosis patients

DETAILED DESCRIPTION:
Until recently, relapsing-remitting multiple sclerosis (RRMS) was considered a homogeneous form of multiple sclerosis (MS). Variability both in the immunopathology of active demyelinating lesions in MS and in response to immunomodulatory treatments has demonstrated that RRMS is a heterogeneous form of MS. An overwhelming number of trials have supported the use of interferon-β (IFN-β) as a first-line immunomodulatory treatment in RRMS. Approximately 30% of IFN-β treated RRMS patients are non-responders (NR) to treatment. Despite vast clinical experience in the use of IFN-β, its mechanisms of action have not been fully clarified. Interleukin-17 (IL-17) is a proinflammatory cytokine that is secreted by a lineage of T cells named Th17 cells. The Th17 chemokine pathways are essential for the development of central nervous system (CNS) autoimmune diseases such as MS. A high IL-17 concentration in the serum. of people with RRMS is associated with nonresponse to IFN-β therapy. Some animal and human studies have shown that IFN-β inhibits the activity of Th17 cells.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 50 years at time of signing informed consent form.
* Relapsing- remitting multiple sclerosis as per the McDonald 2017 criteria, including an MRI brain satisfying the 2017 radiological criteria.
* Kurtzke EDSS step 0.0 - 6.0.
* At the time of screening, being treated with a stable dose of Interferon Beta 1a for at least 6 months.

Exclusion Criteria:

* they had been treated in the last 30 days with methylprednisolone
* they had changed their IFN-β preparation within the last 18 months
* they had other chronic diseases associated with MS
* they had been previously treated with immunosuppressive agents

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Egyptian Relapsing-Remitting Multiple Sclerosis Patients
Sampling Method: Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Correlation between IL17 levels and patients' response to interferon beta 1a as measured by ELISA | Patients were treated with INF B 1a for at least 6 months
  Anti-inflammatory and disease activity biomarkers

SECONDARY OUTCOMES:
Correlation between IL 22 levels and patients' response to interferon beta 1a, measured by ELISA | Patients were treated with INF B 1a for at least 6 months
  Anti-inflammatory and disease activity biomarkers
Correlation between Expanded Disability Status Scale and patients' response to interferon beta 1a | Patients were treated with INF B 1a for at least 6 months
  Determination disability level (0 - 6), The lowest value means that it is best outcome and the highest value is the worst outcome.
Correlation between malondialdehyde levels and patients' response to interferon beta 1a | Patients were treated with INF B 1a for at least 6 months
  oxidative stress biomarkers
Correlation between MRI load and Patients' response to interferon beta 1a | Patients were treated with INF B 1a for at least 6 months
  Determination of T2 lesions
Correlation between body mass index and patients' response to interferon beta 1 a | Patients were treated with INF B 1a for at least 6 months
  Body weight measurement

CONTACTS AND LOCATIONS:
Locations (1):
- Nasser Institute for Research and Treatment, Cairo, Egypt

REFERENCES:
- [Background] Rudick RA, Polman CH. Current approaches to the identification and management of breakthrough disease in patients with multiple sclerosis. Lancet Neurol. 2009 Jun;8(6):545-59. doi: 10.1016/S1474-4422(09)70082-1. PMID 19446274
- [Background] Lucchinetti C, Bruck W, Parisi J, Scheithauer B, Rodriguez M, Lassmann H. Heterogeneity of multiple sclerosis lesions: implications for the pathogenesis of demyelination. Ann Neurol. 2000 Jun;47(6):707-17. doi: 10.1002/1531-8249(200006)47:63.0.co;2-q. PMID 10852536
- [Background] Hesse D, Krakauer M, Lund H, Sondergaard HB, Langkilde A, Ryder LP, Sorensen PS, Sellebjerg F. Breakthrough disease during interferon-[beta] therapy in MS: No signs of impaired biologic response. Neurology. 2010 May 4;74(18):1455-62. doi: 10.1212/WNL.0b013e3181dc1a94. PMID 20439848
- [Background] Axtell RC, Raman C, Steinman L. Interferon-beta exacerbates Th17-mediated inflammatory disease. Trends Immunol. 2011 Jun;32(6):272-7. doi: 10.1016/j.it.2011.03.008. Epub 2011 Apr 29. PMID 21530402
- [Background] Brucklacher-Waldert V, Stuerner K, Kolster M, Wolthausen J, Tolosa E. Phenotypical and functional characterization of T helper 17 cells in multiple sclerosis. Brain. 2009 Dec;132(Pt 12):3329-41. doi: 10.1093/brain/awp289. PMID 19933767